CLINICAL TRIAL: NCT03139331
Title: Phase 1 Study of Pazopanib in Combination With Irinotecan and Temozolomide (PAZIT) for Children and Young Adults With Relapsed or Refractory Sarcoma
Brief Title: PAZIT Study for Children and Young Adults With Relapsed or Refractory Sarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: UCSF Benioff Children's Hospital Oakland (Other); Dana-Farber Cancer Institute (Other); Alex's Lemonade Stand Foundation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 160821; NCI-2017-01929 (Other: NCI Clinical Trials Reporting Program)
Record Dates: First submitted 2017-04-28; First posted 2017-05-03 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Sarcoma; Refractory Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — pazopanib; Irinotecan; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pazopanib, irinotecan, temozolomide (PAZIT) (Experimental): Patients will receive daily oral pazopanib on days 1-21 in a 21-day cycle. This will be combined with intravenous or oral irinotecan and oral temozolomide on days 1-5. Dosing of irinotecan will be from 25 to 37.5 mg/m2/day for IV dosing or from 45 to 67.5 mg/m2/dose for oral dosing and oral temozolomide will be 100 mg/m2/day for dose levels at each assigned dose level. In the absence of disease progression or unacceptable toxicity, patients will receive cycles of therapy repeating every 21 days for a maximum of 12 months on study.
  Interventions: Drug: Pazopanib; Drug: Irinotecan; Drug: Temozolomide

INTERVENTIONS:
Drug: Pazopanib — Pazopanib will be administered orally as a tablet according to an assigned dose level per protocol. A cycle will be defined as 21 days. Drug dosing for the tablet formulation will be determined using a study-specific nomogram.
Drug: Irinotecan — Patients will be given irinotecan at a dose of 25 mg/m2/dose IV on days 1-5 of a 21-day cycle during Cycle 1. In subsequent cycles, irinotecan may be given intravenously at a dose of 25 to 37.5 mg/m2/dose or orally at a dose of 45 to 67.5 mg/m2/dose on days 1-5 of a 21-day cycle.
  Note that some patients enrolled on an earlier protocol version received 50 mg/m2/dose IV on days 1-5 of the first 21-day cycle and then either 50 mg/m2/dose IV or 90 mg/m2/dose orally for subsequent 21-day cycles. This higher dose level is no longer being given to newly enrolled subjects.
Drug: Temozolomide — Temozolomide will be given at a dose of 100 mg/m2/dose orally on days 1-5 of each 21-day cycle.

SUMMARY:
This is the first study to evaluate the safety and clinical activity of the combination of oral pazopanib, intravenous or oral irinotecan, and oral temozolomide in pediatric and young adult patients with relapsed or refractory sarcomas. This study will use a 3 + 3 design for dose escalation (Part 1), followed by an expansion cohort (Part 2) at the recommended phase 2 dose level.

DETAILED DESCRIPTION:
The combination of irinotecan and temozolomide is well-tolerated and provides an active therapy option for heavily pre-treated patients with sarcoma. The toxicity profile and activity level suggest that this combination will provide a useful platform onto which novel compounds may be added. Pazopanib has been shown to demonstrate single-agent activity in sarcomas in the preclinical and clinical settings. Pazopanib has also been shown to have additive or synergistic effects in preclinical models of sarcomas when combined with cytotoxic chemotherapy. Pharmacokinetic studies of pazopanib and irinotecan as well as pharmacodynamic studies of pazopanib to assess anti-angiogenesis will be performed. Exploratory studies to assess non-invasive methods of monitoring tumor response [circulating tumor DNA and functional imaging by positron emission tomography (PET)/magnetic resonance imaging (MRI) will be performed].

ELIGIBILITY:
Inclusion Criteria:

1. Age: Patients must be 6-30 years of age at the time of study enrollment.
2. Body Surface Area: Eligible patients have a body surface area >/= 0.7 m2 AND be able to swallow whole tablets at the time of study enrollment.
3. Diagnosis: Patients must have had histologic verification of one of the malignancies listed below at original diagnosis or at time of relapse.

   * Ewing sarcoma/peripheral primitive neuroectodermal tumor (PNET)
   * Osteosarcoma
   * Rhabdomyosarcoma
   * Non-rhabdomyosarcoma soft tissue sarcoma
   * Desmoplastic small round cell tumor

   Note: Patients with known involvement of the central nervous system (CNS) by malignancy will be included if there is no evidence of active bleeding or intratumoral hemorrhage on radiographic imaging.
4. Disease Status: Patients must have either measurable or evaluable disease
5. Therapeutic Options: Patient's current disease state must be one for which there is not known curative therapy or therapy proven to prolong survival with an acceptable quality of life.
6. Performance Level: Karnofsky >/= 50% for patients > 16 years of age and Lansky >/= 50% for patients </= 16 years of age.

   Note: Neurologic deficits in patients with metastatic CNS tumors must have been relatively stable for a minimum of 1 week prior to study enrollment. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
7. Prior Therapy: Patients must have fully recovered from the acute toxic effects of all prior anti-cancer therapy.

   Myelosuppressive chemotherapy: Patients must not have received myelosuppressive therapy within 2 weeks of enrollment onto this study (6 weeks if prior nitrosourea).

   Hematopoietic growth factors: At least 14 days after the last dose of a long-acting growth factor (e.g. Neulasta) or 7 days for short-acting growth factor. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair.

   Biologic (anti-neoplastic agent): At least 7 days must have passed after the last treatment with a biologic agent. For agents that have known adverse events occurring beyond 7 days from administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair.

   Immunotherapy: At least 4 weeks since the completion of any type of immunotherapy, e.g. tumor vaccines.

   Monoclonal antibodies: >/= 21 days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to Grade </= 1.

   External beam radiation therapy (XRT): >/= 2 weeks must have elapsed for local palliative XRT (small port) and enrollment on study. At least 24 weeks must have elapsed since prior Total Body Irradiation (TBI), radiation to ≥50% of pelvis, or craniospinal radiation; >/= 6 weeks must have elapsed if the patient has received other substantial bone marrow radiation.

   Stem Cell Transplant (SCT): No evidence of active graft-versus-host disease (GVHD) and >/= 2 months must have elapsed since transplant or rescue.

   Prior treatment with pazopanib, irinotecan, temozolomide: Patients may not have previously received pazopanib. However, patients may have received other vascular endothelial growth factor (VEGF) blocking tyrosine kinase inhibitors. Patients must have recovered from any VEGF blocking drug-related toxicity (e.g., proteinuria).

   Patients previously treated with irinotecan and/or temozolomide will be eligible for this study provided they did not progress while receiving one of these agents.
8. Organ Function Requirements:

Adequate Bone Marrow Function defined as:

* Peripheral absolute neutrophil count (ANC) >/= 750/μL
* Platelet count >/= 75,000/μl (transfusion independent, defined as not receiving platelet transfusions within a 7 day period prior to enrollment)
* Hemoglobin >/= 8.0 g/dL; may receive red blood cell (RBC) transfusions

Adequate Renal and Metabolic Function defined as:

* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >/= 70 mL/min/1.73 m2 or
* A serum creatinine based on age/gender per protocol.

The threshold creatinine values in this Table were derived from the Schwartz formula for estimating GFR utilizing child length and stature data published by the Centers for Disease Control and Prevention (CDC).

* Urine protein to creatinine ratio of <1, a urinalysis that is negative for protein, or a 24-hour urine protein level <1000 mg/dL
* No more than Grade 1 abnormalities of potassium, calcium (confirmed by ionized calcium), magnesium, and phosphorus (supplementation allowed).

Adequate Liver Function defined as:

* Total bilirubin </= 1.5 x upper limit of normal (ULN) for age
* Serum glutamate pyruvate transaminase (SGPT)/alanine aminotransferase (ALT) </= 3.0 x ULN (for the purpose of this study, the ULN for SGPT is 45 U/L)
* Serum albumin >/= 2 g/dL
* Must not have active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones, liver metastases or otherwise stable chronic liver disease per investigator assessment).
* No known positivity of hepatitis B surface antigen (HBsAg), or of positive hepatitis C antibody.

Adequate Cardiac Function defined as:

* Shortening fraction of >/= 27% by echocardiogram (while not receiving medications for cardiac function), or
* Ejection fraction of >/= 50% by gated radionuclide study (while not receiving medications for cardiac function).
* Corrected QT interval (QTc) < 480 msec
* Must not have a history of myocardial infarction, severe or unstable angina, peripheral vascular disease or familial QT prolongation.

Adequate Blood Pressure Control defined as: A blood pressure (BP) </= 95% percentile for age, height, and gender. Patients on stable doses of no more than one anti-hypertensive medication, with a baseline BP </= 95% percentile for age, height, and gender will be eligible.

Central Nervous System Function defined as:

* Patients with a known history of seizures must have well-controlled seizures and may not be receiving enzyme-inducing anti-convulsants
* CNS toxicity </= Grade 2.

Adequate pulmonary function defined as:

* No evidence of dyspnea at rest
* No exercise intolerance

Adequate Coagulation defined as: prothrombin time (PT) and partial thromboplastin time (PTT) </= 1.5 x ULN and an international normalized ratio (INR) </= 1.2.

Exclusion Criteria:

1. Pregnancy or Breast-Feeding: Pregnant or breastfeeding women will not be entered on this study due to risks of fetal and teratogenic adverse events as seen in animal/human studies. Negative pregnancy tests must be obtained in girls who are post-menarchal. Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method. The definition of adequate contraception will be based on the judgment of the principal investigator or designated associate. Study drug may also potentially be secreted in milk and therefore breastfeeding women are excluded.
2. Concomitant Medications:

   Corticosteroids: Patients requiring corticosteroids who have not been on a stable or decreasing dose of corticosteroid for the 7 days prior to enrollment are not eligible.

   Investigational Drugs: patients who are currently receiving another investigational drug are not eligible.

   Anti-cancer Agents or Radiation Therapy: Patients who are currently receiving other anti-cancer agents or radiation therapy are not eligible.

   Anti-hypertensive Medications: Patients who are currently receiving more than one anti-hypertensive medication or whose blood pressure is not controlled as defined by protocol are not eligible for study enrollment.

   Anti-coagulation: Patients must not be on therapeutic anti-coagulation. Prophylactic anti-coagulation (i.e., intraluminal heparin) of venous or arterial access devices is allowed.

   Anti-inflammatory and Anti-platelet Agents: Patients currently receiving aspirin, and/or ibuprofen, or other NSAIDs are not eligible.

   Enzyme-inducing Anti-convulsants: Patients who are currently receiving enzyme-inducing anti-convulsants are not eligible.

   CYP3A4 Substrates and Drugs Causing QTc Prolongation: Patients receiving drugs with a known risk of torsades de pointes are not eligible. A list of enzyme inducing, enzyme inhibiting, and other prohibited drugs is provided by the protocol.

   Note: This list includes the prohibition of grapefruit for 14 days prior to enrollment.

   Thyroid Replacement Therapy: Patients who require thyroid replacement therapy are not eligible if they have not been receiving a stable replacement dose for at least 4 weeks prior to study enrollment.
3. Patients who are unable to swallow whole tablets are not eligible.
4. Infection: Patients who have an active or uncontrolled infection are not eligible.
5. Bleeding and Thrombosis: Patients will be excluded if any of the following are present:

   * Evidence of active bleeding, intratumoral hemorrhage, or bleeding diathesis.
   * History (within 6 months prior to study enrollment) of pulmonary embolism, deep vein thrombosis (DVT), or other venous thromboembolic event.
   * History of hemoptysis within 6 weeks prior to study enrollment.
6. Patients with known involvement of the CNS by malignancy will be included if there is no evidence of active bleeding or intratumoral hemorrhage on radiographic imaging.
7. Surgery: Patients who have had or are planning to have the following invasive procedures will be excluded:

   * Major surgical procedures, laparoscopic procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1 therapy. Subcutaneous port placement or central line placement is not considered major surgery, but must be placed greater than 48 hours from planned Day 1 of therapy.
   * Core biopsy within 7 days prior to Day 1 therapy.
   * Fine needle aspirate or central line placement within 48 hours prior to Day 1 therapy.

   Note: Routine bone marrow aspirate and biopsy for the purposes of disease staging are not part of these exclusion guidelines.
8. Patients with serious or non-healing wound, ulcer, or bone fracture.
9. History of abdominal fistula, gastrointestinal perforation, pneumothorax, or intra-abdominal abscess within 28 days of study enrollment.
10. Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible.
11. Patients with history of allergic reactions attributed to compounds of similar composition to pazopanib, irinotecan, or temozolomide are not eligible.

Ages: 6 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 3 weeks
  Maximum tolerated dose or recommended phase 2 dose of pazopanib administered in combination with irinotecan and temozolomide
Number of Patients with Dose-Limiting Toxicities (DLTs) Using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 | 3 weeks
  Toxicity will be graded using the CTCAE criteria, version 4.0. DLT will be defined as any of the events as defined per the protocol that are at least possibly, probably, or definitely attributable to the combination of pazopanib, irinotecan, and temozolomide. DLTs are generally grade 3 or greater in severity.
  Dose limiting hematological and non-hematological toxicities are defined differently, per the protocol.
Describing toxicities of PAZIT drug combination using NCI CTCAE Version 4.0 | 3 weeks
  To describe any toxicities associated with the combination of pazopanib, irinotecan and temozolomide (PAZIT).

SECONDARY OUTCOMES:
Objective Response Rate Using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 | From treatment initiation until disease progression, an average of about 6 months
  The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). The patient's best response assignment will depend on the achievement of both measurement and confirmation criteria. Tumor response will be assessed using RECIST version 1.1.
Progression-Free Survival (PFS) Using RECIST Version 1.1 | From treatment initiation until disease progression, an average of about 6 months
  PFS is defined as the duration of time from start of treatment to time of tumor progression. Tumor response will be assessed using RECIST version 1.1.
Overall Survival (OS) | From treatment initiation until death, an average of about 1 year
  OS is defined as the duration of time from start of treatment to time of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Kieuhoa Vo, MD, MAS, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - UCSF Benioff Children's Hospital, Oakland, Oakland, California
  - University of California, San Francisco, San Francisco, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No